CLINICAL TRIAL: NCT03559803
Title: A Prospective Study of Dynamic Monitoring Specific Immune Response in Locally Advanced Cervix Cancer After Radio-chemotherapy
Brief Title: A Prospective Study of Monitoring Immune Response in Locally Advanced Cervix Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Oncology, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHR-002
Record Dates: First submitted 2018-04-09; First posted 2018-06-18 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; PD-L1; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin (Experimental): Weekly cisplatin (40 mg/m²) will be administered during radiotherapy. At least 3 cycles of cisplatin should be performed according to the hematological and renal functions but not mandatory.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Drug: Cisplatin injection Weekly cisplatin (40 mg/m²) will be administered during radiotherapy. At least 3 cycles of cisplatin should be performed according to the hematological and renal functions but not mandatory.
  Combination Product: radiotherapy A total dose of 45Gy in 25 fractions to the PTV is considered standard but simultaneous integrated boost or two steps boost to specific volumes (positive lymph nodes for example) are accepted and left to the investigator's discretion).
  Other Names: radiotherapy

SUMMARY:
Perspectives:

To analyse if the change of specific immune response will correlate with clinical effect of advanced cervix cancer after radio-chemotherapy.

To evaluate the specific immune response throughout monitor the change of the programmed death-1(PD-1) in CD8 T cell and CD4 T cell and Treg cell in blood at baseline, before first brachytherapy and before the last brachytherapy in the advanced Cervix Cancer patients.

To use immunohistochemistry (IHC) technique to monitor the change of programmed death-ligand 1 (PD-L1),CD68,CD8,CD4,PD1 and Treg expression in biopsy at baseline, before first brachytherapy and before the last brachytherapy in the advanced Cervix Cancer patients.

To detect the change of T cell receptor(TCR) repertoire and Tumor mutation burden (TMB) at baseline, before first brachytherapy and before the last brachytherapy in the advanced Cervix Cancer patients.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common cancer among women worldwide. At present, patients with cervical cancer are treated with radical hysterectomy and pelvic lymphadenectomy or chemoradiation. To improve the prognosis of cervical cancer patients, novel immunotherapeutic strategies need to be developed. Now there are some clinical phase I/II trials ongoing to assess the effects of ipilimumab, pembrolizumab and nivolumab in advanced cervical cancer,but information on the clinical significance of PD-L1 expression in cervical cancer is largely lacking.In this study, the investigator's primary objective:

To analyse if the change of specific immune response will correlate with clinical effect of advanced cervix cancer after radio-chemotherapy.

To evaluate the specific immune response throughout monitor the change of PD-1 in CD8 T cell and CD4 T cell and Treg cell in blood at baseline, before first brachytherapy and before the last brachytherapy in the advanced Cervix Cancer patients.

To use IHC technique to monitor the change of PD-L1, CD68,CD8,CD4,PD1 and Treg expression in biopsy at baseline, before first brachytherapy and before the last brachytherapy in the advanced Cervix Cancer patients.

To detect the change of TCR repertoire and TMB at baseline, before first brachytherapy and before the last brachytherapy in the advanced Cervix Cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-70 years.
2. All FIGO stages cervical cancers which are the matter for radiochemotherapy and exclusive brachytherapy indications.
3. ECOG:0-1.
4. Ability to give informed consent.

4. Patients must be affiliated to a Social Security System. 6. Patient information and written informed consent form signed.

Exclusion Criteria:

1. Known autoimmune disorder.
2. History of HIV and/ or active hepatitis infection.
3. History of pelvic radiation or radio-chemotherapy.
4. Recurrent or metastatic cervical cancer.
5. Contra-indication for cisplatin.
6. Patient pregnant and/or breastfeeding.
7. Patients with psychological or familial disease potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The change of expression of PD-L1+ on cervix biopsies | From baseline,3 weeks,2 months
  The biopsy was collected at baseline,3 weeks,2 months

SECONDARY OUTCOMES:
The change of expression of PD1 on the non-regulatory CD4+ and CD8+ lymphocytes and Treg cells | baseline,3 weeks,2 months
  The blood was collected at baseline,3 weeks,2 months
The diversity of T-cell Repertoire in cervix biopsies and blood, respectively | baseline,3 weeks,2 months
  The blood and biopsies were collected at baseline,3 weeks,2 months
The change of expression of CD8+PD1+ lymphocytes infiltrate on cervix biopsies | baseline,3 weeks,2 months
  The biopsy was collected at baseline,3 weeks,2 months

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - Guizhou Province People's Hospital, Guizhou, Guizhou
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jayshree RS, Sreenivas A, Tessy M, Krishna S. Cell intrinsic & extrinsic factors in cervical carcinogenesis. Indian J Med Res. 2009 Sep;130(3):286-95. PMID 19901438
- [Background] Folkl A, Bienzle D. Structure and function of programmed death (PD) molecules. Vet Immunol Immunopathol. 2010 Mar 15;134(1-2):33-8. doi: 10.1016/j.vetimm.2009.10.006. Epub 2009 Oct 14. PMID 19931186
- [Background] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Background] Yang CY, Lin MW, Chang YL, Wu CT, Yang PC. Programmed cell death-ligand 1 expression in surgically resected stage I pulmonary adenocarcinoma and its correlation with driver mutations and clinical outcomes. Eur J Cancer. 2014 May;50(7):1361-9. doi: 10.1016/j.ejca.2014.01.018. Epub 2014 Feb 15. PMID 24548766
- [Background] Madore J, Vilain RE, Menzies AM, Kakavand H, Wilmott JS, Hyman J, Yearley JH, Kefford RF, Thompson JF, Long GV, Hersey P, Scolyer RA. PD-L1 expression in melanoma shows marked heterogeneity within and between patients: implications for anti-PD-1/PD-L1 clinical trials. Pigment Cell Melanoma Res. 2015 May;28(3):245-53. doi: 10.1111/pcmr.12340. Epub 2014 Dec 22. PMID 25477049
- [Background] Muenst S, Schaerli AR, Gao F, Daster S, Trella E, Droeser RA, Muraro MG, Zajac P, Zanetti R, Gillanders WE, Weber WP, Soysal SD. Expression of programmed death ligand 1 (PD-L1) is associated with poor prognosis in human breast cancer. Breast Cancer Res Treat. 2014 Jul;146(1):15-24. doi: 10.1007/s10549-014-2988-5. Epub 2014 May 20. PMID 24842267
- [Background] Shi F, Shi M, Zeng Z, Qi RZ, Liu ZW, Zhang JY, Yang YP, Tien P, Wang FS. PD-1 and PD-L1 upregulation promotes CD8(+) T-cell apoptosis and postoperative recurrence in hepatocellular carcinoma patients. Int J Cancer. 2011 Feb 15;128(4):887-96. doi: 10.1002/ijc.25397. PMID 20473887
- [Background] Heeren AM, Punt S, Bleeker MC, Gaarenstroom KN, van der Velden J, Kenter GG, de Gruijl TD, Jordanova ES. Prognostic effect of different PD-L1 expression patterns in squamous cell carcinoma and adenocarcinoma of the cervix. Mod Pathol. 2016 Jul;29(7):753-63. doi: 10.1038/modpathol.2016.64. Epub 2016 Apr 8. PMID 27056074
- [Background] Lim SH, Hong M, Ahn S, Choi YL, Kim KM, Oh D, Ahn YC, Jung SH, Ahn MJ, Park K, Zo JI, Shim YM, Sun JM. Changes in tumour expression of programmed death-ligand 1 after neoadjuvant concurrent chemoradiotherapy in patients with squamous oesophageal cancer. Eur J Cancer. 2016 Jan;52:1-9. doi: 10.1016/j.ejca.2015.09.019. Epub 2015 Nov 26. PMID 26623522
- [Background] Zhang J, Fang W, Qin T, Yang Y, Hong S, Liang W, Ma Y, Zhao H, Huang Y, Xue C, Huang P, Hu Z, Zhao Y, Zhang L. Co-expression of PD-1 and PD-L1 predicts poor outcome in nasopharyngeal carcinoma. Med Oncol. 2015 Mar;32(3):86. doi: 10.1007/s12032-015-0501-6. Epub 2015 Feb 22. PMID 25702326